CLINICAL TRIAL: NCT03854344
Title: Prospective Study of Liposomal Bupivacaine for Pain Control of Split Thickness Skin Graft Donor Sites
Brief Title: Liposomal Bupivacaine Versus Lidocaine for Skin Graft Donor Site Pain
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Dhaval Bhavsar, Medical Director Burnett Burn Center, Department of Plastic Surgery Associate Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 143321
Record Dates: First submitted 2019-02-08; First posted 2019-02-26 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Pain, Postoperative; Burns
MeSH Terms: conditions — Pain, Postoperative; Burns | interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Phase 1 -randomized pre-operatively to receive either lidocaine or liposomal bupivicaine Phase 2- all enrolled into regional nerve block group
Who Masked: Participant
Masking Description: Only subjects in first phase will be blinded to their randomization group. Study subject number will be linked to their randomization group. Blinding may be broken if the subject experiences an adverse reaction to the medication utilized for their group so that they are aware that they cannot receive the medication in the future.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): Liposomal Bupivicaine (266mg/20ml) will be diluted into Lactated Ringer solution (280 ml) and injected once intra-operatively subcutaneously before donor site harvesting
  Interventions: Drug: Liposomal bupivacaine
- Group 2 (Active Comparator): Lidocaine (50 mg/50 ml) will be diluted into Lactated Ringer (1000ml) and injected once subcutaneously before donor site harvesting
  Interventions: Drug: Lidocaine Hydrochloride
- Group 3 (Experimental): Subjects will receive regional anesthesia with a bupivacaine nerve block; either a fascia iliaca, lateral femoral cutaneous, or femoral nerve block based on the proposed donor site location
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — Injected subcutaneously for skin graft harvesting
  Arms: Group 2
Drug: Liposomal bupivacaine — Injected subcutaneously for skin graft harvesting
  Other Names: Exparel
  Arms: Group 1
Drug: Bupivacaine Hydrochloride — Used for regional nerve block for skin graft harvesting
  Arms: Group 3

SUMMARY:
Donor site pain study comparing post-operative donor site pain and opioid consumption after use of Lidocaine, Liposomal Bupivicaine or regional nerve block for split thickness skin graft harvesting in patients with less than 20% TBSA burn wounds and less than %5 Deep partial or full thickness burn wounds.

DETAILED DESCRIPTION:
The first phase of the study was a randomized controlled study. In the second phase, all subjects will receive fascia iliaca, lateral femoral cutaneous, or femoral nerve blocks based on the proposed donor site location and will be compared to historic controls from the first phase. In the first phase, the control group underwent split thickness autografting using the standard protocol, involving injection of lidocaine with epinephrine at the donor site. In the first phase, the experimental group underwent injection of liposomal bupivacaine (Exparel) at the time of harvest of the skin graft. In the second phase, patients will undergo preoperative regional anesthesia with a fascia iliaca, lateral femoral cutaneous, or femoral nerve block based on the proposed donor site location rather than the standard protocol of lidocaine with epinephrine at the donor site. Thus, in the second phase, group 3 (preoperative block group) will be compared to historic controls which received the standard of care in the first phase of this trial. Baseline pain levels will be obtained for all subjects using a validated pain assessment scale, the Visual Analog Pain Scale. Postoperatively, time to first opioid pain medication (excluding immediate postoperative recovery from anesthesia), total opioid consumption on a daily basis, and donor site interval pain scores using a validated pain assessment scale will be obtained. The experimental groups will then be individually compared to the control group to determine if there is a significant difference in pain levels, time to first opioid, and overall opioid consumption between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Spanish/English speaking
* <20%TBSA; <5% TBSA deep partial or full thickness burns

Exclusion Criteria:

* chronic pain syndrome
* > 20% TBSA burn injury; > 5% TBSA deep partial or full thickness burn
* pregnant
* allergy to lidocaine or other local anesthetics
* burns to anterior thighs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
A measurement of post operative pain involving skin graft donor site using visual analog scale (VAS) ranging 0-10, at 8 hours post-operatively | The subject completes a pain assessment at 8 hours post-operatively.
  Pain score involving skin graft donor sites are measured using a Visual Analog Scale, which is a horizontal line numbered 0-10, with 10 being the worst pain imaginable and 0 indicating no pain and compare pain scores between donor sites treated with Exparel Vs Lidocaine

SECONDARY OUTCOMES:
Opioid pain medication consumption up to 72 hours post-operatively will be compared between the subjects who are given liposomal bupivacaine (Exparel) and lidocaine at the donor sites | 72 hours (3 days) post operatively
  Opioid consumption will be measured by converting all opioids given to subjects to morphine equivalents
Pain Scores over 72 hours after surgery | Pain scores associated with skin graft donor site will be assessed using Visual Analog Scale (0-10) at 4,8, 12, 24, 48 and 72 hours after surgery. They will be compared between two groups.
  Pain score involving skin graft donor sites are measured using a Visual Analog Scale, which is a horizontal line numbered 0-10, with 10 being the worst pain imaginable and 0 indicating no pain and compare pain scores between donor sites treated with Exparel Vs Lidocaine

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Kansas Health System, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Egan KG, Guest R, Sinik LM, Nazir N, De Ruyter M, Ponnuru S, Bhavsar D. Evaluation of Liposomal Bupivacaine at Split-Thickness Skin Graft Donor Sites Through a Randomized, Controlled Trial. J Burn Care Res. 2021 Nov 24;42(6):1280-1285. doi: 10.1093/jbcr/irab129. PMID 34216466

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/44/NCT03854344/Prot_SAP_000.pdf